CLINICAL TRIAL: NCT05768724
Title: Beneficial Effects of Resemena Diet on Anthropometric, Metabolic and Reproductive Profile in Adolescents With Obesity and Polycystic Ovary Syndrome: a Randomized Controlled Intervention Study
Brief Title: Two Different Dietary Interventions for Girls With Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Esra Döğer, Principal Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Gazi University Medicine
Record Dates: First submitted 2023-02-22; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Polycystic Ovary Syndrome; Obesity; Androgen; Hypersecretion; Diet, Healthy
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity

STUDY DESIGN:
Intervention Model Description: single-blind, randomized, two-arm, parallel six-month dietary intervention.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All cases were assigned codes. The codes were sealed in opaque envelops and kept in statistician ofce until the last patient completed the study.Study personnel involved in the analysis of the results (endocrinologist, radiologist, nurse, and laboratory technicians) were blinded to group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention group (Experimental): METAbolic Syndrome REduction in NAvarra (RESMENA) diet was applied to adolescents with PCOS
  Interventions: Behavioral: intervention diet
- conrol group (Experimental): American Heart Association (AHA) guidelines based diet was applied to adolescents with PCOS
  Interventions: Behavioral: control diet

INTERVENTIONS:
Behavioral: intervention diet — The Resmena diet: It was characterized by a higher meal frequency, consisting of seven meals/d (including breakfast, lunch, dinner, and two snacks in the morning and two snacks in the afternoon), and by a different macronutrient distribution; 40% total energy value from CHO, 30% from proteins and 30% from lipids. This pattern tried to reinforce high n-3 polyunsaturated FA (n-3 PUFA) and high natural antioxidant food consumption and promoted low GL CHO intake as well as a high adherence to the Mediterranean diet. It also maintained a healthy FA profile and a cholesterol content of less than 300 mg/day.
  * Daily meal plans were created according to the energy intake of the participants and sent to the participants via social media every week. Participants were asked to keep 3-day diet records to evaluate their compliance with the diet and were invited to the research center once a month to be checked.
  Arms: İntervention group
Behavioral: control diet — Control diet: It was based on the American Heart Association (AHA) guidelines, including 3-5 meals per day, a macronutrient distribution of 55% total energy value from carbohydrates, 15% proteins, and 30% lipids, a healthy fatty acids (FA) profile and a cholesterol consumption lower than 300 mg/day.
  - Daily meal plans were created according to the energy intake of the participants and sent to the participants via social media every week. Participants were asked to keep 3-day diet records to evaluate their compliance with the diet and were invited to the research center once a month to be checked
  Arms: conrol group

SUMMARY:
This study was conducted to evaluate the efficacy of the MEtabolic Syndrome REduction in NAvarra (RESMENA) diet versus a control diet based on American Heart Association (AHA) recommendations for the treatment of PCOS in adolescents with obesity and PCOS. A total of 40 adolescents diagnosed with PCOS between the ages of 13-18 years were randomized to either a Resmena or control diet for 6 months. Dietary status, anthropometry, body composition, biochemical parameters, and reproductive endocrine hormones were compared between the 2 groups before and after the intervention.

DETAILED DESCRIPTION:
The purpose of this study was to investigate the effect of a high meal frequency, low carbohydrate, high protein, high n-3 PUFA, healthy fatty acid and antioxidant content, low glycemic load Resmena diet or a control diet based on AHA recommendations on anthropometric measurements, body composition, insulin resistance, lipid metabolism levels, inflammatory markers and reproductive endocrine levels in adolescents with obesity and PCOS..Randomized controlled study design was used in the study. Patients in the study were allocated to the control and study intervention groups. Participants were invited to face-to-face interviews at the beginning of the study and monthly for 6 months.

Anthropometric measurements, body composition analysis, and a physical activity questionnaire were performed at the beginning and end of the study, and three-day food consumption records and blood samples for the measurement of biochemical parameters were collected. In addition, the physical activity and food consumption records of the participants were repeated in monthly controls and their anthropometric measurements and body composition were analyzed and compared.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PCOS in adolescent girls according to the Rotterdam criteria
* Age 13-18 years,
* Body mass index (BMI) ≥ 95th percentile

Exclusion Criteria:

* Other endocrine etiological disorders (Cushing's syndrome, congenital adrenal hyperplasia, McCune Albright syndrome, mutations in the glucocorticoid receptor gene, ovarian and adrenal androgen-secreting tumors, hyperprolactinemia, diabetes mellitus, thyroid dysfunction, adrenal, and other endocrine disorders),
* Cardiovascular and cerebrovascular diseases,
* Hematologic disorders
* Liver and kidney failure
* Mental disorders
* Eating disorders
* Contraceptive use in the last 3 months
* Use of insulin-sensitizing agents
* Use of drugs affecting lipid metabolism (such as fish oil)
* Smoking.

Ages: 13 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — adolescent girls with obesity and PCOS
Enrollment: 40 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-05 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Luteinizing hormone (LH) (IU/L) | change between the first day and the sixth month of the study
  Participants' serum LH levels was determined.
Follicle-stimulating hormone (FSH) (IU/L) | change between the first day and the sixth month of the study
  Participants' serum FSH levels was determined.
Total and free (ng/mL) | change between the first day and the sixth month of the study
  Participants' serum FSH levels was determined.
Prolactin (ng/mL) | change between the first day and the sixth month of the study
  Participants' serum prolactin levels was determined.
Dehydroepiandrosterone sulfate (DHEA-S) (µg/dL) | change between the first day and the sixth month of the study
  Participants' serum DHEA-S levels was determined.
Androstenedione (ng/mL) | change between the first day and the sixth month of the study
  Participants' serum androstenedione was determined.
17-hydroxyprogesterone (17-OH progesterone) (ng/mL) | change between the first day and the sixth month of the study
  Participants' serum 17-OH progesterone was determined.
Sex hormone binding globulin (SHGB) (nmol/L) | change between the first day and the sixth month of the study
  Participants' serum SHGB was determined.
Free Androgen Index (FAI) | change between the first day and the sixth month of the study
  Free Androgen Index (FAI) was calculated according to the equation FAI = [(Total testosterone/ SHBG) × 100]
The Ferriman-Gallwey score (FGS) | change between the first day and the sixth month of the study
  The Ferriman-Gallwey score (FGS) was used to evaluate hirsutism.
fasting blood glucose (mg/dl) | change between the first day and the sixth month of the study
  Participants' fasting blood gucose was calculated.
fasting insulin (IU/ml) | change between the first day and the sixth month of the study
  Participants' fasting insulin was calculated.
HOMA-IR index | change between the first day and the sixth month of the study
  Participants' HOMA-IR index value was calculated using the "fasting blood glucose (mmol/L) x fasting insulin (μU/mL)/22.5" formula
QUICKI index | change between the first day and the sixth month of the study
  Participants' QUICKI index was calculated using the 1/[log(fasting insulin in μU/ml)+log(fasting glucose in mg/dl)].

SECONDARY OUTCOMES:
Total cholesterol (mg/dl) composition | change between the first day and the sixth month of the study
  Participants' serum total cholesterol was determined.
high-density lipoprotein (HDL-C) (mg/dl) | change between the first day and the sixth month of the study
  Participants' serum HDL-C was determined.
low-density lipoprotein (LDL) (mg/dl) | change between the first day and the sixth month of the study
  Participants' serum LDL-C was determined.
triglyceride (mg/dl) | change between the first day and the sixth month of the study
  Participants' serum triglyceride was determined.
high-sensitivity CRP (HsCRP)(mg/l) | change between the first day and the sixth month of the study
  Participants' serum HsCRP was determined.
tumor necrosis factor-alpha (TNF-α) (pg/ml) | change between the first day and the sixth month of the study
  Participants' serum TNF-α determined.
interleukin-6 (IL-6) (pg/ml) | change between the first day and the sixth month of the study
  Participants' serum IL-6 determined.
Weight in kilograms | change between the first day and the sixth month of the study
  Body weight measurement was made.
Height in meters | change between the first day and the sixth month of the study
  Height was measured
BMI = body mass index (kg/m2) | change between the first day and the sixth month of the study
  BMI = [body weight (kg)/(height [m])2]' was calculated
Neck circumference in cm | change between the first day and the sixth month of the study
  Neck circumference was measured
. Waist circumference in cm | change between the first day and the sixth month of the study
  waist circumference was measured
body composition analysis | change between the first day and the sixth month of the study
  body composition analysis (fat mass /kg), fat percentage (%), fat-free mass (kg)) were made by using the InBody 720 (1-1000 kHz; InBody Co., Ltd. Korea)

CONTACTS AND LOCATIONS:
Overall Officials: Rukiye BOZBULUT, Dr, Study Chair — Gazi Univeristy; Mahmut Orhun Çamurdan, prof, Study Chair — Gazi University; Aysun Bideci, prof, Study Director — Gazi University
Locations (1):
- Esra Döğer, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No